CLINICAL TRIAL: NCT04403009
Title: The Clinical Difference Between the Nonfatal Coronavirus Disease 2019 (COVID-19) Patients and the Fatal Cases With Severe COVID-19
Brief Title: The Clinical Difference Between the Nonfatal Patients and the Fatal Patients With Severe COVID-19
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: YLS2020(112)
Record Dates: First submitted 2020-04-21; First posted 2020-05-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus Disease 2019; Character of the Severe Patients
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the nonsevere Coronavirus Disease 2019 Patients
  Interventions: Other: no intervention
- the severe Coronavirus Disease 2019 Patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To investigate the difference of the difference between the nonfatal Coronavirus Disease 2019 (COVID-19) Patients and the fatal Patients .The cross sectional study was undertaken to compare the clinical information (laboratory and radiologic characteristics)of nonfatal participants and fatal cases. The investigators wish figure out the clinical character of the fatal participants. The result may help the physician to find the fatal patients with COVID-19 more easily. The fatal patients with COVID-19 could be treated early.

ELIGIBILITY:
Inclusion Criteria:

* The patients with Coronavirus Disease 2019
* Positive result on real-time reverse-transcriptase-polymerase-chain-reaction
* Positive result on chest computed tomography

Exclusion Criteria:

* No

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with Coronavirus Disease 2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Lymphocyte cell | 2 month
  the counting of Lymphocyte(counts/L)
d-dimer | 2 month
  d-dimer（mg/L）
PLT | 2 month
  the counting of Platelets（(counts/L)）
CRP | 2 month
  the level of C-reactive protein (mg/uL)
LDH | 2 month
  lactate dehydrogenase ( U/L)
CK | 2 month
  creatine kinase (U/L)
PT | 2 month
  prothrombin time(second)
ALT | 2 month
  alanine aminotransferase(U/L)
AST | 2 month
  aspartate aminotransferase(U/L)
NK cell | 2 month
  natural killer cell(counts/L)
PCT | 2 month
  procalcitonin（ng/ml）
IL-6 | 2 month
  interleukin-6(mg/L)

SECONDARY OUTCOMES:
the clinical difference of radiologic characteristics between the fatal patients with COVID -19 and the non fatal cases | 2 months
  CT scan feature

OTHER OUTCOMES:
SPO2 | 2 month
  oxygen Saturation

CONTACTS AND LOCATIONS:
Overall Officials: jianheng zhang, MD, Principal Investigator — First Afiliated hospital of Guangzhou medical university
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong
  - Hankou Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided